CLINICAL TRIAL: NCT07159425
Title: Estimation of Analgetic Effect and Cooperability of Pediatric Patients During Application of Gaseous Mixture of Oxygen:Nitrogen Suboxide 50%:50% for Minimal Invasive Procedures
Brief Title: Estimation of Analgetic Effect and Cooperability of Pediatric Patients During Application of Gass Mixture of Oxygen:Nitrogen Suboxide 50%:50% for Minimal Invasive Procedures
Status: Enrolling by invitation | Type: Observational
Sponsor: Mother and Child Health Institute of Serbia Dr Vukan Cupic (Other)
Responsible Party: Principal Investigator, Ana Mandras, Principal Investigator, Mother and Child Health Institute of Serbia Dr Vukan Cupic
Other Study IDs: 8/154
Record Dates: First submitted 2025-04-12; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Pain; Anxiety; Sedation
Keywords: pain; anxiety; nitrous oxyde; children
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Peditric patients planned for minimal invasive procedure: Patients who will be sedated using oxygen:nitrogen suboxide 50%:50% gas mixture for minimal invasive procedure

SUMMARY:
The goal of this observational study is to observe analgetic and anxiolytic effect of gass mixture of oxygen:nitrigen suboxide 50%:50% in pediatric patients sujected to minimal invasive procedures. The main question it aims to answer is: Does gass mixture of oxygen:nitrigen suboxide 50%:50% has effective anxyolitic and analgetic properties for minimal inavsive procedures in pediatric patients?

ELIGIBILITY:
Inclusion Criteria:

* 1 Age 1-16 years 2 Veinpuncture 3 Arterial line placement 4 Nasogastric tube placement 5 Urinary catheter placement 6 Removal of thoracic drain 7 Skin suture

Exclusion Criteria:

1. Age <1 year or > 16 years
2. Pneumothorax
3. Pneumoperitoneum
4. Pneumocephalus
5. Otitis media
6. Obstructive lung disease
7. Upper airway infection
8. Methylenetetrahydrofolate reductase (MTHF) deficiency
9. Vitamin B12 deficiency
10. Megaloblastic anemia

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: single tertiray center random-sample cohort of pediatric patients undergoing any in-hospital minor invasive procedure during a continuous 12 months period of recruitment.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-01-03 (Estimated); Study Completion 2026-01-03 (Estimated)

PRIMARY OUTCOMES:
Pain score for children from 1 to 4 years | 5 minutes during the minimal invasive procedure
  Pain assessed using pain scale: 1-4 years using FLAAC (Face, Leg, Activity, Cry and Consolability) pain scale. Pain was categorized as: 0-no pain, 1-3 mild, 4-6 moderate and 7-10 severe
Pain score for children from 4 to 9 years. | 5 minutes during the minimal invasive procedure
  Pain assessed using pain scale: 4-9 years using Wong-Baker Faces Pain Rating Scale. Pain was categorized as: 0-no pain, 1-3 mild, 4-6 moderate and 7-10 severe
Pain score for children from 9 to 16 years | 5 minutes during the minimal invasive procedure
  Pain assessed using pain scale: from 9-16 years using Numeric Rating Scale (NRS) Pain was categorized as: 0-no pain, 1-3 mild, 4-6 moderate and 7-10 severe.

SECONDARY OUTCOMES:
anxiolytic effect | 5 minutes during the minimal invasive procedure
  anxiolytic effect qualified as "cooperative" and "uncooperative"
hypotension | measured 5 minutes after initiating application of gase mixture of oxygen:nitrogen oxide 50%:50%
  drop in noninvasive blood pressure for more than 20mmHg value for age
bradycardia | measured 5 minutes after initiating application of gase mixture of oxygen:nitrogen oxide 50%:50%
  Drop in heart rate measured as beats per minute according to age
desaturation | measured 5 minutes after initiating application of gase mixture of oxygen:nitrogen oxide 50%:50%
  fall of hemoglobine oxygen saturation measured by pulse oximetry SpO2 belov 94%
level of sedation | Assessment will be made at the beginig of applicati
  Level of sedation will be estimated using Ramsay sedation scale. The Ramsay sedation scale is a well-established monitoring method to determine the level of awareness. Points assigned are : 1-Patient anxious, agitated, or restless; 2- Patient cooperative, oriented, or tranquil; 3- Patient responds to commands only; 4- Brisk response to a light glabellar tap or loud auditory stimulus; 5 -Sluggish response to a light glabellar tap or loud auditory stimulus; 6-No response

CONTACTS AND LOCATIONS:
Overall Officials: Ana Mandras, PhD, Principal Investigator — Institute for mother and child health care
Locations (1):
- Institute for mother and child health care, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
In order to protect individual patients data IPD will not br shared

REFERENCES:
- [Background] Carbajal R, Biran V, Lenclen R, Epaud R, Cimerman P, Thibault P, Annequin D, Gold F, Fauroux B. EMLA cream and nitrous oxide to alleviate pain induced by palivizumab (Synagis) intramuscular injections in infants and young children. Pediatrics. 2008 Jun;121(6):e1591-8. doi: 10.1542/peds.2007-3104. Epub 2008 May 5. PMID 18458035
- [Background] Ekbom K, Jakobsson J, Marcus C. Nitrous oxide inhalation is a safe and effective way to facilitate procedures in paediatric outpatient departments. Arch Dis Child. 2005 Oct;90(10):1073-6. doi: 10.1136/adc.2004.060319. PMID 16177164
- [Background] Zier JL, Liu M. Safety of high-concentration nitrous oxide by nasal mask for pediatric procedural sedation: experience with 7802 cases. Pediatr Emerg Care. 2011 Dec;27(12):1107-12. doi: 10.1097/PEC.0b013e31823aff6d. PMID 22134227
- [Background] Fein D, Avner JR, Khine H. Pattern of pain management during lumbar puncture in children. Pediatr Emerg Care. 2010 May;26(5):357-60. doi: 10.1097/PEC.0b013e3181db2026. PMID 20404782
- [Background] Milesi C, Pidoux O, Sabatier E, Badr M, Cambonie G, Picaud JC. Nitrous oxide analgesia for intubating preterm neonates: a pilot study. Acta Paediatr. 2006 Sep;95(9):1104-8. doi: 10.1080/08035250600698818. PMID 16938758

DOCUMENTS (1):
  • Study Protocol (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT07159425/Prot_000.pdf